CLINICAL TRIAL: NCT02721680
Title: Refinement and Validation of a Military Emotional Intelligence Training Program
Brief Title: Refinement and Validation of an Awareness Training Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: William D. Killgore (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, William D. Killgore, Principal Investigator, University of Arizona
Organization: University of Arizona (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 1607696724
Record Dates: First submitted 2016-03-01; First posted 2016-03-29 (Estimated); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Awareness Training

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- Healthy Subjects- Awareness Training Group 1 (Experimental): Subjects in this arm will undergo an internal awareness training program.
  Interventions: Other: Internal Awareness Training Program
- Healthy Subjects - Awareness Training Group 2 (Experimental): Subjects in this arm will undergo an external awareness training program.
  Interventions: Other: External Awareness Training Program

INTERVENTIONS:
Other: Internal Awareness Training Program
  Arms: Healthy Subjects- Awareness Training Group 1
Other: External Awareness Training Program
  Arms: Healthy Subjects - Awareness Training Group 2

SUMMARY:
The goal of the proposed project is to provide the Army with a brief, well-validated, internet-based training program for enhancing Awareness Training and resilience skills. This project will address the needs outlined for the Military Operational Medicine Research Program, particularly with regard to enhancing Psychological Health and Resilience. The fundamental approach of the project directly addresses the need to "develop psychological resilience among Service members and families to promote well-being and prevent behavioral health outcomes." Addressing this need is crucial, as military personnel are often required to serve under dangerous and emotionally stressful conditions. Prolonged stress or exposure to very intense life threatening experiences, such as those encountered in combat or other hazardous duty deployments can increase the risk of developing mental health problems including depression, anxiety, or post-traumatic stress disorder (PTSD). One possible way to minimize the effects of these stressful experiences on Service members is to strengthen their emotional flexibility, adaptability, and capacity to cope with adversity before they find themselves faced with such situations. To fill this need, the investigators propose to provide the military with a web-based program that focuses on enhancing Awareness Training, a core set of trainable awareness skills that collectively include the capacity to understand, perceive, control, and use emotions effectively.

While the previous pilot program was successful in some ways, it needs further research before it is ready for widespread use. The investigators therefore propose to build upon the existing strengths already in the program and redesign the weaker modules to be more effective. Over the course of a four-year study, the investigators propose to develop this program. The proposed Awareness Training program is brief, web-based, easily accessible, and sufficiently focused such that it could be completed by large numbers of military personnel with minimal time burden, leading to rapid enhancement of awareness skills. Such a program could have a significant effect in promoting resilience, interpersonal functioning, and brain health among Service members and their families, while reducing the likelihood of mental health problems among those returning from exposure to potentially traumatic experiences.

The central hypothesis is that a set of well designed and targeted training modules addressing core awareness ability domains will significantly enhance measured awareness skills, will translate into improved performance on militarily relevant metrics, and will lead to better mental and emotional health, as well as well being during stressful situations and subsequent cognitive processing.

ELIGIBILITY:
Inclusion Criteria:

* English as a primary language

Exclusion Criteria:

* History of neurological illness, current DSM-5 Axis I disorder
* Traumatic brain injury with loss of consciousness greater than 30 minutes

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1266 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2021-11 (Actual); Study Completion 2021-11 (Actual)

PRIMARY OUTCOMES:
Change in Mayer-Salovey Caruso Emotional Intelligence Test (MSCEIT) | Measured before and after the Awareness Training Program is given on Day 1

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Arizona Psychiatry Department, Tucson, Arizona
  - University of Arizona, Tucson, Arizona